CLINICAL TRIAL: NCT04681508
Title: Myocardial Injury After Non-cardiac Surgery (MINS), Acute Kidney Injury (AKI) and Pulmonary Pathology in Patients Undergoing Acute Abdominal Surgery
Brief Title: MINS, AKI and Pulmonary Pathology in Patients Undergoing Acute Abdominal Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AHA
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Abdomen, Acute; Myocardial Injury; Acute Kidney Injury; Pulmonary Disease
MeSH Terms: conditions — Abdomen, Acute; Acute Kidney Injury; Lung Diseases | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients undergo chest CT without contrast enhancement and chest X-ray. Blood and urine sampling from patients subsequently undergoing emergency laparoscopy or laparotomy. Otherwise standard care
  Interventions: Diagnostic Test: Chest CT without contrast enhancement and chest X-ray

INTERVENTIONS:
Diagnostic Test: Chest CT without contrast enhancement and chest X-ray — Chest CT without contrast enhancement and chest X-ray as supplement to diagnostic abdominal CT

SUMMARY:
Explorative study to investigate potential predictors of myocardial injury, acute kidney injury and pulmonary disorder after acute high-risk abdominal surgery.

DETAILED DESCRIPTION:
The main issues are:

* To investigate if coronary calcification predisposes the development of myocardial injury and causes an increased mortality rate.
* To evaluate the predictive value of NT-pro-BNP in relation to the development of MINS and the mortality rate.
* To evaluate the predictive value of different biomarkers of AKI in relation to which patients develop AKI.
* To examine the proteins, exosomes and single cell RNA during acute kidney injury in order to describe the molecular processes in the kidney during AKI.
* To examine whether a chest CT scan without contrast enhancement will change treatment decisions in the acute gastrointestinal patient compared with a chest x-ray.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Patients included in the AHA regimen undergoing CT on suspicion acute high-risk abdominal disorder e.g.g bowel obstruction GI perforation or ischemia, and need of emergency abdominal surgery, either laparoscopic surgery or laparotomy.
* Able to speak Danish. In case Danish was not spoken an interpreter was used to obtain the informed consent.
* Able to give informed consent.

Exclusion Criteria:

* Patients who cannot give informed consent to participate in the study 15 minutes after receiving verbal information regarding the study.
* Known chronic kidney disease requiring dialysis at the time of admission (only exclusion criteria for the part of the study relating to AKI).
* Patients included in the AHA regimen, but conservative treatment is chosen (only exclusion criteria for the part of the study relating to MINS and AKI).
* Patients not resident in Denmark.
* Patients not able to give informed consent.
* Patient not able to speak Danish and not enough time to obtain an interpreter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with myocardial injury af non-cardiac surgery | 30 days
  Troponin-I above specified level and dynamic changes
Mortality rate | 30 days
  Postoperative mortality
Mortality rate | 90 days
  Postoperative mortality
Mortality rate | 1 year
  Postoperative mortality
Acute kidney Injury | 30 days
  According to KIDGO criteria
Proportion of patients with pulmonary pathology | 1 day
  Findings (including incidental) on a chest x-ray and chest CT scan without contrast enhancement
Proportion of patients with pulmonary complications | 30 days
  Postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, PhD, Study Chair — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No